CLINICAL TRIAL: NCT02247466
Title: Optimizing Surgical Conditions During Laparoscopic Umbilical, Incisional -and Linea Alba Herniotomy With Deep Neuromuscular Blockade
Brief Title: Optimizing Surgical Conditions During Laparoscopic Herniotomy With Deep Neuromuscular Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Roar Medici, MD, research assistant, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NMBDKHernia2014
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Laparoscopic Herniotomy
Keywords: Neuromuscular Blockade; Laparoscopy
MeSH Terms: interventions — Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A - Saline, assesment, rocuronium and assesment (Active Comparator): Intervention after intubation and placement of trocars without NMB. Bolus of saline (placebo) 6mL (TOF 100%) the surgeon assesses the surgical workspace with pneumoperitoneum 12 mmHg. After administration of rocuronium 0.6 mg/kg when TOF=0 the surgical workspace is assessed again
  Interventions: Drug: Rocuronium and Sugammadex
- Group B - Rocuronium, assesment, sugammadex and assesment (Active Comparator): Intervention after intubation and placement of trocars without NMB. Bolus of rocuronium 0.6 mg/kg when TOF=0 the surgeon assesses the surgical workspace with pneumoperitoneum 12 mmHg. Three minutes after administration of sugammadex (TOF 100%) the surgical workspace is assessed again
  Interventions: Drug: Rocuronium and Sugammadex

INTERVENTIONS:
Drug: Rocuronium and Sugammadex

SUMMARY:
The purpose of this study is to investigate surgical work space and surgical conditions in patients scheduled for laparoscopic umbilical, -linea alba and incisional herniotomy. The patients will act as their own control with evaluation of surgical work space and surgical conditions during both deep NMB and no NMB.

DETAILED DESCRIPTION:
Umbilical herniotomy is a frequent surgical procedure worldwide, and the larger hernia defects are preferably operated by laparoscopic technique. The advantages of the laparoscopic approach are shorter convalescence with earlier mobilization, and less wound complications [1]. A preferred approach is currently to close the defect by laparoscopic suturing in order to reduce the formation of seroma in the hernia sac [2] , and then apply a mesh by intraperitoneal onlay technique (IPOM technique). However, it may be difficult to suture the defect if there is tension in the abdominal wall muscles together with the applied pneumoperitoneum.

There is evidence that muscle relaxation improves conditions for endotracheal intubation[3] and reduces laryngeal morbidity but only a few studies investigate the necessity of relaxation during laparoscopic surgery [4].

During laparoscopic surgery muscle relaxation is used with great variability. Sometimes the procedure is performed without muscle relaxation and sometimes with a so-called surgical neuromuscular blockade, which with objective neuromuscular monitoring means that train-of-four (TOF) is kept at 3-4 responses to nerve stimulation of the ulnar nerve. In this way there is a great variability in the neuromuscular blockade and rarely the patients are receiving deep neuromuscular blockade.

Traditionally, neuromuscular monitoring is done by measuring the muscle strength of the adductor pollicis muscle on the thumb. The response to TOF nerve stimulation may be zero, while muscle relaxation of more resistant muscles such as the abdominal muscles and the diaphragm [5;6] are not complete which means that the patients may cough and their abdominal wall may feel "tight" during surgery, even though no response at the thumb is recorded. It is possible to quantify a deep neuromuscular block by the use of post-tetanic-count (PTC). With establishment of deep, continuous neuromuscular blockade with PTC value 0-1 all muscles including abdominal muscles and diaphragm are paralyzed [7]. It is therefore possible, that a deep neuromuscular blockade (NMB) where the diaphragm and the abdominal wall muscles are more paralyzed will optimize the surgical work space, ease the surgical procedure, reduce operative time for the suturing part of the procedure as well as the total procedure time, and reduce the number of recurrences by long term follow-up.

The purpose of this study is to investigate surgical work space and surgical conditions in patients scheduled for laparoscopic umbilical, -linea alba and incisional herniotomy. The patients will act as their own control with evaluation of surgical work space and surgical conditions during both deep NMB and no NMB.

Hypothesis:

Deep NMB defined as TOF=0 and post-tetanic count PTC ≥1, will give better surgical workspace, better surgical conditions, as well as shorter duration of surgery and reduced number of recurrences of hernias compared with no NMB.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Elective laparoscopic umbilical herniotomy, incisional herniotomy and linea alba - herniotomy
* Can read and understand Danish
* Informed consent

Exclusion Criteria:

* Known allergy to sugammadex, rocuronium or mivacurium
* Known homozygous variants in the butyrylcholinesterase gene
* Severe renal disease, defined by S-creatinine> 0.200 mmol/L, GFR < 30ml/min or hemodialysis)
* Neuromuscular disease that may interfere with neuromuscular data
* Lactating or pregnant (Women of child bearing potential must take a urine pregnancy test at the day of the operation. The test will be provided by the hospital staff).
* Indication for rapid sequence induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Ring Gätke, MD, Ph.D., Study Chair — Department of Anaesthesiology, Herlev Hospital
Locations (2):
- Denmark (2):
  - Gentofte Hospital, Hellerup, Capital Region
  - Herlev Hospital, Herlev, Capital Region

REFERENCES:
- [Derived] Soderstrom CM, Borregaard Medici R, Assadzadeh S, Folsgaard S, Rosenberg J, Gatke MR, Madsen MV. Deep neuromuscular blockade and surgical conditions during laparoscopic ventral hernia repair: A randomised, blinded study. Eur J Anaesthesiol. 2018 Nov;35(11):876-882. doi: 10.1097/EJA.0000000000000833. PMID 29878947
- [Derived] Medici R, Madsen MV, Asadzadeh S, Folsgaard S, Rosenberg J, Gatke MR. Neuromuscular blockade during laparoscopic ventral herniotomy: protocol for a randomised controlled trial. Dan Med J. 2015 Aug;62(8):A5120. PMID 26239595

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - Saline, Assesment, Rocuronium and Assesment: Intervention after intubation and placement of trocars without NMB. Bolus of saline (placebo) 6mL (TOF 100%) the surgeon assesses the surgical workspace with pneumoperitoneum 12 mmHg. After administration of rocuronium 0.6 mg/kg when TOF=0 the surgical workspace is assessed again
  Rocuronium and Sugammadex
- Group B - Rocuronium, Assesment, Sugammadex and Assesment: Intervention after intubation and placement of trocars without NMB. Bolus of rocuronium 0.6 mg/kg when TOF=0 the surgeon assesses the surgical workspace with pneumoperitoneum 12 mmHg. Three minutes after administration of sugammadex (TOF 100%) the surgical workspace is assessed again
  Rocuronium and Sugammadex
Period: Overall Study
Arm/Group | Group A - Saline, Assesment, Rocuronium and Assesment | Group B - Rocuronium, Assesment, Sugammadex and Assesment
Started | 19 | 18
Completed | 19 | 15
Not Completed | 0 | 3
Not completed — Procedure changed to open surgery | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Saline, Assesment, Rocuronium and Assesment | Group B - Rocuronium, Assesment, Sugammadex and Assesment | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (17) | 55 (15) | 56.4 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 15 | 10 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index
  kg/m2 | 28 (4) | 30 (4) | 29 (4.17)
ASA 1/2/3 [Count of Participants; unit: Participants] — american society of anesthesiologists Physical Status Classification System score.
  American Society of Anesthesiologists (ASA) Score is a global score that assesses the physical status of patients before surgery.
  It is sometimed refereed to as ASA-PS, because it is a measure of 'physical status'.
  ASA 1 A normal healthy patient. ASA 2 A patient with mild systemic disease. ASA 3 A patient with severe systemic disease. ASA 4 A patient with severe systemic disease that is a constant threat to life. ASA 5 A moribund patient who is not expected to survive
  Participants
    ASA 1 | 5 | 4 | 9
    ASA 2 | 12 | 10 | 22
    ASA 3 | 2 | 1 | 3
Previous abdominal surgery [Count of Participants; unit: Participants] | 12 | 10 | 22
Herniea size (cm) [Mean (Standard Deviation); unit: cm] | 2.4 (1.5) | 3.1 (2.1) | 2.72 (1.82)

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Surgical Workspace
Description: Improvement of surgical workspace (rated on a 5-point scale) estimated as the difference between the workspace during deep NMB and the workspace without NMB. Ratings are performed in the same patient during stable pneumoperitoneum at 12 mmHg.
  (1 Extremely poor conditions; 2 Poor conditions; 3 Acceptable conditions; 4 Good conditions; 5 Optimal conditions)
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Saline, Assesment, Rocuronium and Assesment | Group B - Rocuronium, Assesment, Sugammadex and Assesment
Number analyzed (Participants) | 19 | 15
Participants
  Changes in ratings 5 to 3 | 0 | 1
  Changes in ratings 4 to 3 | 0 | 0
  Changes in ratings 5 to 4 | 0 | 4
  Changes in ratings 3 to 3 | 1 | 0
  Changes in ratings 4 to 4 | 1 | 2
  Changes in ratings 5 to 5 | 14 | 4
  Changes in ratings 4 to 5 | 2 | 2
  Changes in ratings 3 to 4 | 0 | 1
  Changes in ratings 3 to 5 | 1 | 1

2. Secondary Outcome: Surgical Conditions While Suturing
Description: Surgeon´s rating of surgical conditions while suturing the hernia (5-point rating scale)
  (1 Extremely poor conditions; 2 Poor conditions; 3 Acceptable conditions; 4 Good conditions; 5 Optimal conditions)
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Saline, Assesment, Rocuronium and Assesment | Group B - Rocuronium, Assesment, Sugammadex and Assesment
Number analyzed (Participants) | 19 | 13
Participants
  1. Extremely poor conditions | 0 | 0
  2. Poor conditions | 0 | 0
  3. Acceptable conditions | 0 | 2
  4. Good conditions | 3 | 4
  5. Optimal conditions | 16 | 7

3. Secondary Outcome: Operating Time
Description: Duration of operating time (from first incision to last suture)
Time Frame: 3 hours
Measure: Mean (Full Range); unit: minutes
Arm/Group | Group A - Saline, Assesment, Rocuronium and Assesment | Group B - Rocuronium, Assesment, Sugammadex and Assesment
Number analyzed (Participants) | 19 | 15
minutes | 61 [37 to 85] | 64 [33 to 95]

4. Secondary Outcome: Suturing Time
Description: Duration of suturing the hernia (minutes)
Time Frame: 3 hours
Measure: Mean (Full Range); unit: minutes
Arm/Group | Group A - Saline, Assesment, Rocuronium and Assesment | Group B - Rocuronium, Assesment, Sugammadex and Assesment
Number analyzed (Participants) | 19 | 15
minutes | 10 [1 to 19] | 9 [2 to 16]

5. Secondary Outcome: Contractions
Description: Sudden contractions of the abdominal wall during operation (bucking or coughing), number of participants with sudden contractions
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Saline, Assesment, Rocuronium and Assesment | Group B - Rocuronium, Assesment, Sugammadex and Assesment
Number analyzed (Participants) | 19 | 15
Participants | 1 | 0

6. Secondary Outcome: Insufflator Alarms
Description: Insufflator alarms where pneumoperitoneum > 17 mmHg Number of patients experiencing insufflator alarms where pneumoperitoneum > 17 mmHg
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Saline, Assesment, Rocuronium and Assesment | Group B - Rocuronium, Assesment, Sugammadex and Assesment
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

7. Secondary Outcome: Continuous Abdominal Contractions
Description: Number of patients experiencing episodes with continuous abdominal contractions where the abdomen feels "tight" but the operation can still proceed (the intestines are gradually displaced near the inner surface of the abdominal wall)
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Saline, Assesment, Rocuronium and Assesment | Group B - Rocuronium, Assesment, Sugammadex and Assesment
Number analyzed (Participants) | 19 | 15
Participants | 0 | 0

8. Secondary Outcome: Recurrences of Hernias
Description: Number of recurrences of hernias by 2 year follow-up (separate publication).
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Patients will be observed during their stay at the hospital and will be contacted by telephone on first and seventh postoperative day. Possibly adverse events during this period will be reported. Finally the patient´s case files will be reviewed for reports of adverse events at 17-21 days after operation.
Arm/Group | Group A - Saline, Assesment, Rocuronium and Assesment | Group B - Rocuronium, Assesment, Sugammadex and Assesment
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT02247466/Prot_SAP_000.pdf